CLINICAL TRIAL: NCT03668782
Title: Efficacy of Umbilical Cord Milking in Elective Cesarean Section
Brief Title: Cord Milking in Elective Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Policlinico Abano Terme (Other)
Responsible Party: Principal Investigator, Vincenzo Zanardo, Director of Perinatal Medicine, Policlinico Abano Terme
Other Study IDs: 24/2018 Fondazione Leonardo
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Placental Transfusion
MeSH Terms: conditions — Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After the infant was delivered, the obstetrician either immediately clamped and cut the cord or initiated the milking protocol intervention, near the cord insertion site on the placenta towards the infant, three times before clamping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- immediate cord clamping: Tthe umbilical cord of neonates was cut and clamped.
  Interventions: Procedure: Umbilical cord milking
- umbilical cord milking.: Tthe umbilical cord of neonates was milked.
  Interventions: Procedure: Umbilical cord milking

INTERVENTIONS:
Procedure: Umbilical cord milking — The babies were held at the level of the placenta, while the umbilical cord was milked or cut and clamped.
  Other Names: Immediate cord clamping

SUMMARY:
The objective of the study was to investigate the efficacy and safety of umbilical cord milking as compared with immediate cord clamping on placental transfusion, estimated by Δ hematocrit between cord blood at birth and capillary heel hematocrit at 48 hours of age, in elective cesarean delivered neonates.

ELIGIBILITY:
Inclusion Criteria: singleton low risk pregnancy, gestational age of 39 to 40/0 weeks confirmed by a first trimester ultrasound, no evidence of active labor, 18 years of age, and (5) a written consent given by the woman.

-

Exclusion Criteria:maternal medical and obstetric complications, severe anemia, clotting disorders and suspected intrauterine growth restriction

-

Ages: 1 Minute to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All women who presented for an elective cesarean section were screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Placental transfusion | 48 hours
  Δ hematocrit between cord blood at birth and capillary heel hematocrit at 48 hours of age

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Abano Terme, Abano Terme, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zanardo V, Guerrini P, Severino L, Simbi A, Parotto M, Straface G. A Randomized Controlled Trial of Intact Cord Milking versus Immediate Cord Clamping in Term Infants Born by Elective Cesarean Section. Am J Perinatol. 2021 Mar;38(4):392-397. doi: 10.1055/s-0039-1697673. Epub 2019 Oct 10. PMID 31600796